CLINICAL TRIAL: NCT05075915
Title: Transfusion and COVID-19
Acronym: TRANSCOV-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7958
Record Dates: First submitted 2021-10-11; First posted 2021-10-13 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; Blood donation; Blood transfusion; Labile products; Blood platelets; Psoralen; ECMO; SARS-CoV-2; Consumption of blood products
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alsace was particularly and early on affected by SARS-CoV-2 and quickly implemented a reduction in scheduled admissions and non-urgent surgical interventions, making it possible to reduce requests for labile blood products linked to non-urgent surgical procedures. as has been reported in the literature; the population containment measures also led to a major reduction in traffic - and consequently accidents on the public roads. At the same time, other demands for blood products related to activities such as onco-hematology were little affected. Finally, the blood banks have adapted their collection procedure.

To answer these questions, we propose to conduct a retrospective study over two parallel periods of 2019 and 2020 of the consumption of blood products on the one hand and the availability of stocks on the other hand.

ELIGIBILITY:
Inclusion criteria:

* Adults patient (≥18 years old)
* Patients admitted to Strasbourg University Hospitals for suspicion of Covid-19, between February 24 and May 31 of 2019 and 2020
* Labile blood products consumed between February 24 and May 31 of 2019 and 2020
* Subjects not having his opposition, after information, to the reuse of his data for the purposes of this research.

Non-inclusion criteria:

* Patients who expressed opposition to participating in the study
* Patients under legal protection
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) admitted to Strasbourg University Hospitals for suspicion of Covid-19, between February 24 and May 31 of 2019 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Study of the consumption of labile blood products at Strasbourg University Hospitals, during the two covid-19 periods: from February 24 to May 31, 2019 and 2020 | Files analysed retrospectively from from February 24 to May 31, 2019 and from February 24 to May 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Michel MERTES, MD, PhD, Principal Investigator — Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'Anesthésie et Réanimation chirurgicale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France